CLINICAL TRIAL: NCT06025461
Title: Correlation Between Multi-modal Ultrasound Features and Pathologic Classification of BI-RADS Category 4 Breast Lesions
Brief Title: Multimodal Ultrasound Diagnosis Characteristics of Bi-rads Class 4 Breast Lesions
Status: Completed | Type: Observational
Sponsor: Ma Zhe (Other)
Responsible Party: Sponsor-Investigator, Ma Zhe, Director of Ultrasound, Qianfoshan Hospital
Organization: Qianfoshan Hospital (Other)
Other Study IDs: YXLL-KY-2023(012)
Record Dates: First submitted 2023-08-30; First posted 2023-09-06 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-08

CONDITIONS: Breast Disease
MeSH Terms: conditions — Breast Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- fibroadenoma group
  Interventions: Other: no intervention
- breast hyperplasia group
  Interventions: Other: no intervention
- other types of benign nodules group
  Interventions: Other: no intervention
- non-specific invasive carcinoma group
  Interventions: Other: no intervention
- other types of breast cancer group
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
Objective: To explore the potential association between the multimodal ultrasound characteristics and pathological classification of BI-RADS category 4 breast lesions, so as to clarify the diagnostic characteristics of multimodal ultrasound in different pathological types BI-RADS category 4 breast lesions.

Materials and methods: Patients who visited in The First Affiliated Hospital of Shandong First Medical University ＆ Shandong Provincial Qianfoshan Hospital were collected. Their general clinical features, information on preoperative ultrasound diagnosis, and postoperative pathologic data were reviewed.

ELIGIBILITY:
Inclusion Criteria:

* Perform ultrasound examination at our hospital before surgery or puncture biopsy; Complete histopathological data; Two ultrasound physicians with more than 5 years of experience in breast ultrasound diagnosis were diagnosed as BI-RADS Class 4 based on preoperative ultrasound images.

Exclusion Criteria:

* Poor image quality; Incomplete clinical data.

Ages: 30 Years to 76 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who visited in The First Affiliated Hospital of Shandong First Medical University ＆ Shandong Provincial Qianfoshan Hospital were collected.
Sampling Method: Probability Sample
Enrollment: 85 (Actual)
Dates: Start 2021-11-15 (Actual); Primary Completion 2023-03-30 (Actual); Study Completion 2023-03-30 (Actual)

PRIMARY OUTCOMES:
elasticity imaging/B-mode ratio | Immediately record the elastic modulus value after the patient receives routine ultrasound and shear wave elastography
  The ratio of lesion length on strain elastography images to lesion length on grayscale images
shear wave velocity | Immediately record the elastic modulus value after the patient receives routine ultrasound and shear wave elastography
  Shear wave velocity values at the hardest point of the lesion and surrounding tissues
strain ratio | Immediately record the elastic modulus value after the patient receives routine ultrasound and shear wave elastography
  The ratio of average strain between surrounding tissues at the same depth and the lesion

CONTACTS AND LOCATIONS:
Locations (1):
- QianfoshanH, Shandong, China

IPD SHARING:
Plan to Share IPD: No